CLINICAL TRIAL: NCT05004883
Title: Targeting Food Cue Responsiveness for Weight Loss
Brief Title: Solutions for Hunger and Regulating Eating
Acronym: SHARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Minnesota (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Kerri Boutelle, Ph.D., Professor, Herbert Wertheim School of Public Health and Longevity Science and School of Medicine Departments of Pediatrics and Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201362; R01DK122504 (NIH)
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
Keywords: Food Responsiveness; Satiety Responsiveness; Weight Loss; Overeating
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Hyperphagia | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Regulation of Cues Enhanced Treatment (Experimental): The ROC program provides psychoeducation, coping skills, self-monitoring and experiential learning, and it will be combined with aspects of BWL to capitalize on the strengths of both treatments.
  Interventions: Behavioral: Regulation of Cues Enhanced
- Behavioral Weight Loss (Active Comparator): The BWL program will include dietary recommendations, physical activity recommendations, and behavioral change recommendations.
  Interventions: Behavioral: Behavioral Weight Loss
- Nutrition, Stress Management, and Social Support (Active Comparator): Nutrition Education, Stress Management and Social Support will be covered. Mindfulness will be practiced in every session.
  Interventions: Behavioral: Nutrition Education, Stress Management and Social Support

INTERVENTIONS:
Behavioral: Regulation of Cues Enhanced — ROC is based on the Behavioral Susceptibility Theory and designed to incorporate psychoeducation, cue-exposure treatment, appetite awareness training, coping skills, and self-monitoring of satiety and cravings to treat high Food Responsiveness and low Satiety Responsiveness. BWL and ROC will be integrated for this arm, to capitalize on the strengths of both treatments. All participants will be taught to decrease caloric intake and increase physical activity, and to use all of the behavioral skills provided in BWL. However, they will also be taught models of hunger and satiety and about food cue reactivity, and will learn skills to manage these. This arm will include an experiential component, including hunger monitoring during dinner and participating in exposure exercises.
  Other Names: ROC+
  Arms: Regulation of Cues Enhanced Treatment
Behavioral: Behavioral Weight Loss — The BWL program includes dietary, physical activity, and behavioral change recommendations. All participants will be instructed on how to consume a balanced deficit diet of conventional foods; individual goals for energy intake will be based on initial body weight. Participants will be instructed in measuring portion sizes, counting calories, and self-monitoring food intake. The physical activity program will focus on increasing both lifestyle activity and structured exercise programs. Behavior change recommendations include stimulus control, self-monitoring, goal setting, managing high-risk situations, meal planning, slowing eating, problem solving, social support, cognitive restructuring, lapse and relapse prevention skills, and maintaining weight loss.
  Other Names: BWL
  Arms: Behavioral Weight Loss
Behavioral: Nutrition Education, Stress Management and Social Support — Topics included will be stress management/relaxation, social support, and nutrition education. There will be a strong mindfulness component to this group.
  Arms: Nutrition, Stress Management, and Social Support

SUMMARY:
The objective of this proposed study is to collect efficacy data on ROC+ compared to an active comparator (AC) and to Behavioral Weight Loss (BWL) for participants who are high in Food Responsiveness.

DETAILED DESCRIPTION:
The investigators have developed a new model for the treatment of obesity, called Regulation of Cues (ROC), which is based on Behavioral Susceptibility Theory. The ROC program targets two theorized mechanisms for overeating; decreased sensitivity to appetitive cues and increased sensitivity to external food cues. Considering that BWL has merit for some people, but fails to facilitate maintenance, this study will compare BWL, ROC with some aspects of BWL (ROC+) and an active comparator (AC). All treatment groups will be 1.5 hours (including weigh-ins) and will be provided in groups of 15-20 participants weekly for 4 months and twice a month for 2 months (total treatment duration = 6 months, 20 meetings). The investigators will recruit adults with overweight or obesity who are high in Food Responsiveness (FR) and will assess them at baseline, post-treatment (month 6), mid-follow-up (month 12) and follow-up (month 18).

ELIGIBILITY:
Inclusion Criteria:

* high Food Responsiveness
* BMI between 25kg/m^2 and 45kg/m^2
* able to read English at a 5th grade reading level
* willing and able to participate in assessment visits and treatment sessions, whether held in-person or via password protected Zoom meetings
* able to provide data through questionnaires
* has a smart phone through which they can complete Ecological Momentary Assessments

Exclusion Criteria:

* major medical conditions such as diabetes or recent history of coronary heart disease; symptoms of angina, stroke, osteoarthritis, osteoporosis, orthopedic problems that would limit activity during the following 18 months; or any other serious medical condition that would make physical activity unsafe
* bulimia or anorexia, significant cognitive impairment, a known psychotic disorder, acute suicidal ideation, moderate or severe alcohol or substance use disorder, or unstable psychiatric illness (e.g., recent psychiatric hospitalization in the past year)
* medical or psychological problems that could make adherence with the study protocol difficult or dangerous
* pregnant, lactating, or planning to become pregnant in the next 18 months
* participating in other weight control programs and/or taking medication for weight loss
* previous bariatric surgery
* moving out of the San Diego area for the duration of their study enrollment (18 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index | Change from baseline at an average of 6 months, 9 months, 12 months, 15 months, and 18 months
  Body Mass Index as measured by height and weight

SECONDARY OUTCOMES:
Change in Food Responsiveness As Measured by the FR Scale of the AEBQ | Change from baseline at an average of 6 months, 12 months, and 18 months
  The Adult Eating Behavior Questionnaire (AEBQ) assesses appetitive traits, including food responsiveness, hunger, and satiety responsiveness. We will use the food responsiveness (FR) scale to measure participants' food responsiveness at a given time point. The score for the FR scale ranges from 4-20, with higher scores indicating higher food responsiveness, and lower scores indicating lower food responsiveness.
Change in Satiety Responsiveness As Measured by the SR Scale of the AEBQ | Change from baseline at an average of 6 months, 12 months, and 18 months
  The Adult Eating Behavior Questionnaire (AEBQ) assesses appetitive traits, including food responsiveness, hunger, and satiety responsiveness. We will use the satiety responsiveness (SR) scale to measure participants' satiety responsiveness at a given time point. The score for the SR scale ranges from 4-20, with higher scores indicating higher satiety responsiveness, and lower scores indicating lower satiety responsiveness.
Change in Inhibition As Measured by the Stop Signal Task | Change from baseline at an average of 6 months, 12 months, and 18 months
  Go stimuli are four pictures of food in landscape or portrait format; participants must respond to the go stimuli by pressing the left and right response keys on the keyboard. On 25% of trials, a visual stop signal will be presented; participants are instructed to withhold responding when this signal is presented. This task measures inhibitory control.
Change in Restriction As Measured by the TFEQ | Change from baseline at an average of 6 months, 12 months, and 18 months
  The Three-Factor Eating Questionnaire (TFEQ) assesses three cognitive and behavioral domains of eating: cognitive restraint, disinhibition, and hunger. We will use the restraint subscale to measure restriction. Scores on the restraint subscale range from 0-21, with lower scores indicating less restriction and higher scores indicating more restriction.
Change in Caloric Intake As Measured by the DHQ III | Change from baseline at an average of 6 months, 12 months, and 18 months
  The Diet History Questionnaire III consists of 135 food and beverage line items and 26 dietary supplement questions. Some line items for foods and beverages have additional embedded questions that allow for final assignment to items in the nutrient and food group database leading to 263 foods/beverages listed in the database. For example, a single line item asks frequency of intake and portion size of soda or soft drinks. Embedded underneath are questions regarding whether the soft drinks consumed are regular vs. diet or caffeinated vs. decaffeinated. Answers to these questions lead to assignment of one of four food codes in the database: diet soda with caffeine, diet soda without caffeine, regular soda with caffeine or regular soda without caffeine. We will use this to measure caloric intake.
Change in Eating Cognitions As Measured by the FCQ-T-reduced | Change from baseline at an average of 6 months, 12 months, and 18 months
  The shortened version of the Food Craving Questionnaire - Trait (FCQ-T-reduced) assesses food cravings and evaluates food craving traits. We will use it to measure eating cognitions. Item scores range from 1-6, and the overall score ranges from 15-90, with higher scores indicating with more food craving cognitions, and lower scores indicating fewer food craving cognitions.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States

REFERENCES:
- [Derived] Boutelle KN, Eichen DM, Obayashi S, Pasquale EK, Strong DR, Tietz AS, Reed KL, Peterson CB. Design of the SHARE study: A randomized controlled trial evaluating the regulation of cues treatment for adults with overweight or obesity and high food responsiveness. Contemp Clin Trials. 2025 Aug;155:107970. doi: 10.1016/j.cct.2025.107970. Epub 2025 Jun 1. PMID 40460908